CLINICAL TRIAL: NCT02641912
Title: A Clinical Study to Evaluate the Efficacy of an Experimental Mouthwash Formulation
Brief Title: Potential of an Experimental Mouthwash Formulation to Reduce Dry Mouth Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 204870
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — Mineral Waters

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Mouthwash (Experimental): During supervised product use: Participants will rinse with 15 mls of mouthwash for 30 seconds and spit out. No rinsing with water immediately after product usage is permitted. At Home use:Participants will rinse with 15 mls of mouthwash for 30 seconds and spit out. A maximum of two doses can be used per day.
  Interventions: Other: Biotene mouthwash
- Mineral Water (Other): During supervised product use:Participants will take a dose (drink) of one measured sip of 15mls of water.
  At Home use: Participants can sip (drink) water as often as required. Participants will be consuming their own water for home use.
  Interventions: Other: Mineral Water

INTERVENTIONS:
Other: Biotene mouthwash — During supervised product use: Participants will rinse with 15 mls of mouthwash for 30 seconds and spit out. No rinsing with water immediately after product usage is permitted. At Home use:Participants will rinse with 15 mls of mouthwash for 30 seconds and spit out. A maximum of two doses can be used per day.
  Arms: Experimental Mouthwash
Other: Mineral Water — During supervised product use:Participants will take a dose (drink) of one measured sip of 15mls of water.
  At Home use: Participants can sip (drink) water as often as required. Participants will be consuming their own water for home use.
  Arms: Mineral Water

SUMMARY:
This will be a single center, 7-day, examiner blind, two treatment-arm, randomized, stratified (Sjogren's Syndrome status [Y/N]), parallel group study conducted in participants experiencing dry mouth symptoms. This study is designed to investigate the effect of an experimental mouthwash formulation in providing relief of dry mouth symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon oral examination
* Subject with stable and controlled condition with no overt medical conditions which would contraindicate participation (in the opinion of the Investigator or medically qualified designee) and no clinically significant and relevant abnormalities of medical history or oral examination which would interfere with the conduct of the study
* All subjects should report having a feeling of a dry mouth according to the DMSQ. (Subject must answer at least 2 out of the 4 questions with 'agree a little', 'agree' or 'strongly agree'
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 14 days of the screening visit
* Previous participation in this study
* Recent history (within the last 1 year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family
* Subjects with Sjögren's Syndrome along with reporting having a feeling of dry mouth according to the DMSQ, should also have a confirmed diagnosis of their condition as shown by a positive salivary gland biopsy or SS-A (anti-Ro antibody) or SS-B (La antibody) or a letter from a physician if diagnosis was made more than 3 years ago OR Subjects reporting having a feeling of dry mouth due to other diseases or conditions excluding Sjögren's Syndrome
* Understands and is willing, able and likely to comply with all study procedures and restrictions.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Subject is currently undergoing radiotherapy and/or chemotherapy treatment
* Any condition the investigator identifies that can confound the subject's ability to properly participate in the study e.g. Alzheimer's Disease
* Subjects with untreated oral mucosal disease which in the opinion of the investigator could interfere with the study (e.g. current oral ulceration)
* Evidence of gross intra-oral neglect or need for extensive dental therapy

  -. Denture wearer (complete dentures)
* Subjects not on stable doses of prescription systemic parasympathetic medications (e.g. Pilocarpine), for the treatment of the feeling of dry mouth
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 14 days of the screening visit
* Previous participation in this study
* Recent history (within the last 1 year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in United States of America.
Pre-assignment Details: A total of 104 participants were screened. Out of which 100 participants were randomized and stratified based on confirmed Sjögren's syndrome status (Yes[Y]/No[N]).
Groups:
- Experimental Mouthwash: During supervised product use: Participants rinsed with 15 milliliter (mL) of mouthwash for 30 seconds and spat out. No rinsing with water immediately after product usage was permitted. At Home: Participants rinsed with 15 mL of mouthwash for 30 seconds and spat out. A maximum of two doses were used per day.
- Mineral Water: During supervised product use: Participants took a dose (drink) of one measured sip of 15mL of water. At Home: Participants drank water as often as required. Participants consumed their own water for home use.
Period: Overall Study
Arm/Group | Experimental Mouthwash | Mineral Water
Started | 53 | 47
Completed | 53 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Mouthwash: During supervised product use: Participants rinsed with 15 mL of mouthwash for 30 seconds and spat out. No rinsing with water immediately after product usage was permitted. At Home: Participants rinsed with 15 mL of mouthwash for 30 seconds and spat out. A maximum of two doses were used per day.
- Total: Total of all reporting groups
Arm/Group | Experimental Mouthwash | Mineral Water | Total
Number analyzed (Participants) | 53 | 47 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.66 (14.418) | 51.57 (14.111) | 51.09 (14.210)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 64
  Male | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Mean Response to the Question 1 'Relieving the Discomfort of Dry Mouth' in Product Performance and Attributes Questionnaire 3 (PPAQ3) at 120 Minutes(Mins) Post Treatment on Day 8
Description: Participants answered question 1 'Relieving the discomfort of dry mouth' in PPAQ3 and rated this question on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 120 mins post treatment on Day 8
Population: Intent-to-treat (ITT) population which included all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed for this outcome is the part of ITT population for specific question at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 52 | 37
score on a scale | 2.50 (1.057) | 1.89 (1.149)
Statistical Analysis 1: Comparison: Experimental Mouthwash vs Mineral Water; Test type: Superiority or Other; p = 0.0084, ANOVA; From ANOVA model with factors for treatment and confirmed Sjögren's syndrome status stratification using Observed Margins option; Least sqaure (LS) mean difference = 0.63, 95% CI 2-sided [0.17 to 1.10] — Difference is first named treatment minus second named treatment such that a positive difference favours the first named treatment

2. Secondary Outcome: Mean Response to the Question 1 'Relieving the Discomfort of Dry Mouth' in Product Performance And Attributes Questionnaire 2 (PPAQ2) at 30 Mins Post Treatment on Day 8
Description: Participants answered to the question 1 'Relieving the discomfort of dry mouth' in PPAQ2 and rated this question on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 30 mins post treatment on Day 8
Population: ITT population which included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed for this outcome is the part of ITT population for specific question at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 39
score on a scale | 2.92 (1.053) | 2.26 (1.163)

3. Secondary Outcome: Mean Response to the Question 1 'Relieving the Discomfort of Dry Mouth' in PPAQ3 at 60 and 240 Mins Post Treatment on Day 8
Description: Participants answered to the question 1 'Relieving the discomfort of dry mouth' in PPAQ3 and rated this question on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 60 and 240 mins post treatment on Day 8
Population: Analysis for this outcome was conducted on ITT population which included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment of efficacy. n= number of participants analyzed for this outcome for specific question at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  At 60 min. (n= 52, 38) | 2.71 (1.091) | 1.97 (1.197)
  At 240 min. (n=53, 35) | 2.42 (1.151) | 1.77 (1.087)

4. Secondary Outcome: Mean Response to Product Performance And Attributes Questionnaire1(PPAQ1) at 5 Mins Post Treatment on Day 8
Description: Participants answered 3 questions in PPAQ1. Q1= Having a immediate dry mouth relief; Q2= Having a immediate lubricating effect; Q3= Having a immediate moisturizing effect. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 5 mins post treatment on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Having a Immediate Dry Mouth Relief(n=53, 42) | 3.57 (1.169) | 3.02 (1.297)
  Having a Immediate Lubricating Effect(n=53,43) | 3.58 (1.247) | 2.67 (1.304)
  Having a Immediate Moisturizing Effect(n=53,43) | 3.55 (1.234) | 2.93 (1.183)

5. Secondary Outcome: Mean Response to Question(Q) Number 2 to 11 (Q2 to Q11) From PPAQ2 at 30 Mins Post Treatment on Day 8
Description: Participants answered questions, Q2-Q11 in PPAQ2. Q2=Feeling comfortable in the mouth; Q3=Soothing your mouth; Q4= Allowing you to speak without difficulty; Q5= Effectively moistens your mouth; Q6= Effectively lubricates your mouth; Q7= Helping to freshen your breath; Q8= Protecting your mouth from drying out; Q=9 Providing whole mouth comfort; Q10= Helping you to swallow without difficulty; Q11= Helping mouth feel normal. These questions were rated on a scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 30 mins post treatment on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q2: Feeling Comfortable in The Mouth(n=53,39) | 3.00 (1.019) | 2.28 (1.169)
  Q3: Soothing Your Mouth(n=53,38) | 3.02 (1.065) | 2.34 (1.169)
  Q4:Allowing to Speak Without Difficulty(n=46,34) | 3.11 (1.059) | 2.59 (1.184)
  Q5: Effectively Moistens Your Mouth(n= 53,39) | 3.02 (1.101) | 2.33 (1.177)
  Q6: Effectively Lubricates Your Mouth(53,38) | 3.04 (1.091) | 2.24 (1.173)
  Q7: Helping to Freshen Your Breath(n=52,34) | 3.06 (1.162) | 2.18 (1.336)
  Q8: Protecting Your Mouth From Drying Out(53,38) | 2.98 (1.118) | 2.13 (1.070)
  Q9: Providing Whole Mouth Comfort(n=53,39) | 3.02 (1.118) | 2.18 (1.073)
  Q10:Helping to Swallow Without Difficulty(n=49,34) | 3.00 (1.041) | 2.41 (1.184)
  Q11: Helping Mouth Feel 'Normal'(n=53,38) | 2.92 (1.053) | 2.26 (1.107)

6. Secondary Outcome: Mean Response to Question (Q) Number 2 to 14 (Q2-Q14) From PPAQ3 at 60 Mins. Post Treatment on Day 8
Description: Participants answered Q2- Q14 from PPAQ3. Q2= Feeling comfortable in the mouth; Q3= Soothing your mouth; Q4= Allowing you to speak without difficulty; Q5= Effectively moistens your mouth; Q6= Effectively lubricates your mouth; Q7= Helping to freshen your breath; Q8= Protecting your mouth from drying out; Q9= Providing whole mouth comfort; Q10= Helping you to swallow without difficulty; Q11= Helping mouth feel normal; Q12= Having a long lasting dry mouth relief; Q13= Having a long lasting lubricating effect; Q14= Having a long lasting moisturizing effect. These question were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 60 mins. post treatment on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q2: Feeling Comfortable in The Mouth(n=53,39) | 2.77 (1.086) | 2.03 (1.203)
  Q3: Soothing Your Mouth(n=52,36) | 2.79 (1.109) | 1.92 (1.180)
  Q4:Allowing to Speak Without Difficulty(n=46,34) | 2.96 (1.154) | 2.44 (1.284)
  Q5: Effectively Moistens Your Mouth(n= 53,37) | 2.79 (1.166) | 1.95 (1.177)
  Q6: Effectively Lubricates Your Mouth(52,38) | 2.83 (1.133) | 1.95 (1.184)
  Q7: Helping to Freshen Your Breath(n=52,32) | 2.75 (1.135) | 1.94 (1.318)
  Q8:Protecting Your Mouth From Drying Out(n=53,38) | 2.77 (1.120) | 2.00 (1.252)
  Q9: Providing Whole Mouth Comfort(n=53,38) | 2.75 (1.108) | 1.95 (1.207)
  Q10:Helping to Swallow Without Difficulty(n=48,32) | 2.81 (1.065) | 2.22 (1.289)
  Q11: Helping Mouth Feel 'Normal'(n=53,38) | 2.77 (1.137) | 1.97 (1.197)
  Q12:Having Long Lasting Dry Mouth Relief(n=53,38) | 2.72 (1.116) | 1.82 (1.182)
  Q13:Long Lasting Lubricating Effect(n=53,36) | 2.75 (1.175) | 1.72 (1.137)
  Q14:Long Lasting Moisturizing Effect(n=53,36) | 2.74 (1.163) | 1.78 (1.174)

7. Secondary Outcome: Mean Response to Question (Q) Number 2 to 14 (Q2-Q14) From PPAQ3 at 120 Mins. Post Treatment on Day 8
Description: as for outcome 6
Time Frame: 120 mins. post treatment on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q2: Feeling Comfortable in The Mouth(n=53,39) | 2.58 (1.117) | 1.90 (1.095)
  Q3: Soothing Your Mouth(n=53,39) | 2.57 (1.152) | 1.85 (1.089)
  Q4:Allowing to Speak Without Difficulty(n=45,34) | 2.67 (1.087) | 2.26 (1.189)
  Q5: Effectively Moistens Your Mouth(n= 53,39) | 2.60 (1.115) | 1.77 (1.087)
  Q6: Effectively Lubricates Your Mouth(53,38) | 2.64 (1.194) | 1.74 (1.107)
  Q7: Helping to Freshen Your Breath(n=52,33) | 2.44 (1.195) | 1.82 (1.236)
  Q8: Protecting Your Mouth From Drying Out(53,38) | 2.49 (1.137) | 1.79 (1.143)
  Q9: Providing Whole Mouth Comfort(n=52,36) | 2.54 (1.111) | 1.86 (1.175)
  Q10:Helping to Swallow Without Difficulty(n=49,34) | 2.63 (1.112) | 2.03 (1.167)
  Q11: Helping Mouth Feel 'Normal'(n=53,38) | 2.64 (1.128) | 1.89 (1.085)
  Q12:Having Long Lasting Dry Mouth Relief(n=53,37) | 2.57 (1.233) | 1.68 (0.973)
  Q13:Long Lasting Lubricating Effect(n=53,37) | 2.57 (1.201) | 1.73 (1.071)
  Q14:Long Lasting Moisturizing Effect(n=53,36) | 2.57 (1.169) | 1.75 (1.052)

8. Secondary Outcome: Mean Response to Questions (Q) Number 2 to 14 (Q2 to Q14) From PPAQ3 at 240 Mins. Post Treatment on Day 8
Description: as for outcome 6
Time Frame: 240 mins. post treatment on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q2: Feeling Comfortable in The Mouth(n=53,37) | 2.47 (1.154) | 1.81 (1.101)
  Q3: Soothing Your Mouth(n=53,37) | 2.40 (1.182) | 1.68 (1.002)
  Q4:Allowing to Speak Without Difficulty(n=46,32) | 2.70 (1.113) | 2.13 (1.212)
  Q5: Effectively Moistens Your Mouth(n= 53,37) | 2.45 (1.202) | 1.73 (1.071)
  Q6: Effectively Lubricates Your Mouth(53,36) | 2.45 (1.218) | 1.78 (1.098)
  Q7: Helping to Freshen Your Breath(n=51,31) | 2.45 (1.189) | 1.74 (1.182)
  Q8: Protecting Your Mouth From Drying Out(53,37) | 2.43 (1.201) | 1.68 (1.056)
  Q9: Providing Whole Mouth Comfort(n=53,37) | 2.43 (1.135) | 1.73 (1.018)
  Q10:Helping to Swallow Without Difficulty(n=48,32) | 2.63 (1.214) | 1.88 (1.129)
  Q11: Helping Mouth Feel 'Normal'(n=53,36) | 2.38 (1.147) | 1.78 (1.098)
  Q12:Having Long Lasting Dry Mouth Relief(n=53,37) | 2.36 (1.145) | 1.76 (1.140)
  Q13:Long Lasting Lubricating Effect(n=53,37) | 2.34 (1.192) | 1.65 (1.086)
  Q14:Long Lasting Moisturizing Effect(n=53,37) | 2.40 (1.182) | 1.65 (1.086)

9. Secondary Outcome: Mean Response to Product Performance And Attributes Questionnaire 4(PPAQ4) Prior to Treatment on Day 8
Description: Participants answered the 9 questions of PPAQ4. Q1= Providing relief all night; Q2= Reducing the number of times you wake up from dry mouth; Q3= Feeling less parched when you wake up; Q4= Having a long lasting dry mouth relief; Q5= Having a long lasting lubricating effect; Q6= Having a long lasting moisturizing effect; Q7= Having an overall dry mouth relief; Q8= Having an overall lubrication effect; Q9= Having an overall moisturizing effect. These question were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: prior to treatment on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Providing Relief All Night(n=47,31) | 2.68 (1.163) | 1.71 (1.160)
  Reducing Number of Wake Up from Dry Mouth(n=41,27) | 2.80 (1.209) | 1.81 (1.272)
  Feeling Less Parched When You Wake Up(n=47,32) | 2.51 (1.196) | 1.84 (1.110)
  Having a Long Lasting Dry Mouth Relief(n=47,32) | 2.68 (1.270) | 1.75 (0.950)
  Having a Long Lasting Lubricating Effect(n=49,33) | 2.63 (1.253) | 1.70 (0.918)
  Having a Long Lasting Moisturizing Effect(n=48,31) | 2.69 (1.257) | 1.65 (0.915)
  Having an Overall Dry Mouth Relief(n=49,34) | 2.73 (1.132) | 1.76 (1.017)
  Having an Overall Lubrication Effect(n=49,32) | 2.63 (1.202) | 1.78 (0.975)
  Having an Overall Moisturizing Effect(n=49,33) | 2.67 (1.197) | 1.70 (0.984)

10. Secondary Outcome: Mean Response to PPAQ1 at 5 Mins Post Treatment on Day 1
Description: Participants answered to the 3 question in PPAQ1. Q1= Having a immediate dry mouth relief; Q2= Having a immediate lubricating effect; Q3= Having a immediate moisturizing effect. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 5 mins post treatment on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Having a Immediate Dry Mouth Relief(n=51,45) | 3.55 (0.986) | 3.11 (1.402)
  Having a Immediate Lubricating Effect(n=53,43) | 3.43 (0.971) | 3.02 (1.371)
  Having a Immediate Moisturizing Effect(n=53,45) | 3.57 (1.029) | 3.38 (1.211)

11. Secondary Outcome: Mean Response to PPAQ2 at 30 Mins Post Treatment on Day 1
Description: Participants answered to the 11 question in PPAQ2. Q1= Relieving the discomfort of dry mouth; Q2= Feeling comfortable in the mouth; Q3= Soothing your mouth; Q4= Allowing you to speak without difficulty; Q5= Effectively moistens your mouth; Q6= Effectively lubricates your mouth; Q7= Helping to freshen your breath; Q8= Protecting your mouth from drying out; Q9= Providing whole mouth comfort; Q10= Helping you to swallow without difficulty; Q11= Helping mouth feel normal. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 30 mins post treatment on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Mouthwash: During supervised product use: Participants were instructed to rinse their mouth with 15 mL of mouthwash for 30 seconds and spit out. Immediate rinsing with water after product usage was not permitted. At Home use: Participants were instructed to rinse their mouth with 15 mL of mouthwash for 30 seconds and spit out. A maximum of two doses were allowed to use per day.
- Mineral Water: During supervised product use: Participants were instructed to take a dose (drink) of one measured sip of 15mL of water. At Home: Participants were instructed to drink water as often as required. Participants consumed their own water for home use.
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort Of Dry Mouth(n=53,45) | 2.92 (0.958) | 2.33 (1.261)
  Q2:Feeling Comfortable in The Mouth(n=52,45) | 2.92 (0.926) | 2.36 (1.151)
  Q3:Soothing Your Mouth(n=52,45) | 2.94 (0.895) | 2.29 (1.180)
  Q4:Allowing to Speak Without Difficulty(n=46,41) | 3.13 (0.833) | 2.51 (1.075)
  Q5: Effectively Moistens Your Mouth(n= 53,44) | 3.08 (0.997) | 2.41 (1.226)
  Q6: Effectively Lubricates Your Mouth(n=53,45) | 3.06 (0.949) | 2.29 (1.160)
  Q7: Helping to Freshen Your Breath(n=52,38) | 3.21 (0.997) | 2.03 (1.219)
  Q8: Protecting Your Mouth From Drying Out(n=53,43) | 2.92 (0.997) | 2.07 (1.280)
  Q9: Providing Whole Mouth Comfort(n=53,43) | 3.06 (0.949) | 2.35 (1.289)
  Q10:Helping to Swallow Without Difficulty(n=51,43) | 3.06 (0.904) | 2.60 (1.348)
  Q11: Helping Mouth Feel 'Normal'(n=53,44) | 3.02 (0.951) | 2.32 (1.377)

12. Secondary Outcome: Mean Response to PPAQ3 at 60 Mins Post Treatment on Day 1
Description: Participants answered to the 14 questions in PPAQ3. Q1= Relieving the discomfort of dry mouth; Q2= Feeling comfortable in the mouth; Q3= Soothing your mouth; Q4= Allowing you to speak without difficulty; Q5= Effectively moistens your mouth; Q6= Effectively lubricates your mouth; Q7= Helping to freshen your breath; Q8= Protecting your mouth from drying out; Q9= Providing whole mouth comfort; Q10= Helping you to swallow without difficulty; Q11= Helping mouth feel normal; Q12= Having a long lasting dry mouth relief; Q13= Having a long lasting lubricating effect; Q14= Having a long lasting moisturizing effect. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 60 mins post treatment on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort Of Dry Mouth(n=53,40) | 2.60 (1.044) | 2.15 (1.272)
  Q2:Feeling Comfortable in The Mouth(n=53,44) | 2.68 (0.915) | 2.18 (1.167)
  Q3:Soothing Your Mouth(n=52,42) | 2.65 (0.926) | 2.19 (1.234)
  Q4:Allowing to Speak Without Difficulty(n=47,39) | 3.04 (0.955) | 2.59 (1.208)
  Q5: Effectively Moistens Your Mouth(n= 53,43) | 2.79 (1.150) | 2.21 (1.407)
  Q6: Effectively Lubricates Your Mouth(53,41) | 2.70 (1.153) | 2.02 (1.214)
  Q7: Helping to Freshen Your Breath(n=51,38) | 2.86 (1.059) | 1.82 (1.159)
  Q8:Protecting Your Mouth From Drying Out(n=53,41) | 2.49 (1.120) | 2.02 (1.275)
  Q9: Providing Whole Mouth Comfort(n=53,41) | 2.58 (1.027) | 2.17 (1.160)
  Q10:Helping to Swallow Without Difficulty(n=51,40) | 2.65 (1.036) | 2.30 (1.244)
  Q11: Helping Mouth Feel 'Normal'(n=53,43) | 2.62 (1.042) | 2.05 (1.194)
  Q12:Having Long Lasting Dry Mouth Relief(n=53,43) | 2.55 (1.136) | 1.88 (1.219)
  Q13:Long Lasting Lubricating Effect(n=53,41) | 2.57 (1.152) | 1.95 (1.264)
  Q14:Long Lasting Moisturizing Effect(n=53,41) | 2.62 (1.113) | 2.00 (1.245)

13. Secondary Outcome: Mean Response to PPAQ3 at 120 Mins Post Treatment on Day 1
Description: as for outcome 12
Time Frame: 120 mins post treatment on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort Of Dry Mouth(n=52,40) | 2.48 (1.146) | 2.13 (1.324)
  Q2:Feeling Comfortable in The Mouth(n=52,40) | 2.56 (1.145) | 2.10 (1.236)
  Q3:Soothing Your Mouth(n=52,40) | 2.48 (1.075) | 2.13 (1.305)
  Q4:Allowing to Speak Without Difficulty(n=48,40) | 2.75 (1.194) | 2.50 (1.240)
  Q5: Effectively Moistens Your Mouth(n= 52,39) | 2.52 (1.229) | 2.23 (1.441)
  Q6: Effectively Lubricates Your Mouth(52,39) | 2.50 (1.146) | 2.10 (1.294)
  Q7: Helping to Freshen Your Breath(n=51,31) | 2.59 (1.203) | 2.00 (1.265)
  Q8:Protecting Your Mouth From Drying Out(n=53,40) | 2.30 (1.153) | 2.00 (1.281)
  Q9: Providing Whole Mouth Comfort(n=53,39) | 2.45 (1.202) | 2.21 (1.260)
  Q10:Helping to Swallow Without Difficulty(n=52,39) | 2.48 (1.146) | 2.28 (1.317)
  Q11: Helping Mouth Feel 'Normal'(n=52,40) | 2.50 (1.146) | 2.28 (1.261)
  Q12:Having Long Lasting Dry Mouth Relief(n=52,39) | 2.42 (1.194) | 1.97 (1.347)
  Q13:Long Lasting Lubricating Effect(n=53,37) | 2.36 (1.226) | 1.92 (1.211)
  Q14:Long Lasting Moisturizing Effect(n=53,39) | 2.42 (1.167) | 1.95 (1.255)

14. Secondary Outcome: Mean Response to PPAQ3 at 240 Mins Post Treatment on Day 1
Description: Participants answered to the 14 questions in PPAQ3 as follows: Q1= Relieving the discomfort of dry mouth; Q2= Feeling comfortable in the mouth; Q3= Soothing your mouth; Q4= Allowing you to speak without difficulty; Q5= Effectively moistens your mouth; Q6= Effectively lubricates your mouth; Q7= Helping to freshen your breath; Q8= Protecting your mouth from drying out; Q9= Providing whole mouth comfort; Q10= Helping you to swallow without difficulty; Q11= Helping mouth feel normal; Q12= Having a long lasting dry mouth relief; Q13= Having a long lasting lubricating effect; Q14= Having a long lasting moisturizing effect. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 240 mins post treatment on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Mouthwash: During supervised product use: Participants rinsed with 15 mL of mouthwash for 30 seconds and spit out. No rinsing with water immediately after product usage was permitted. At Home: Participants rinsed with 15 mL of mouthwash for 30 seconds and spit out. A maximum of two doses were used per day.
- Mineral Water: During supervised product use: Participants took a dose (drink) of one measured sip of 15mL of water. At Home: Participants drunken water as often as required. Participants consumed their own water for home use.
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort Of Dry Mouth(n=53,37) | 2.38 (1.060) | 2.03 (1.213)
  Q2:Feeling Comfortable in The Mouth(n=53,39) | 2.49 (1.137) | 2.08 (1.156)
  Q3:Soothing Your Mouth(n=52,40) | 2.52 (1.146) | 2.08 (1.163)
  Q4:Allowing to Speak Without Difficulty(n=47,35) | 2.60 (1.116) | 2.51 (1.222)
  Q5: Effectively Moistens Your Mouth(n= 52,40) | 2.48 (1.196) | 2.00 (1.132)
  Q6: Effectively Lubricates Your Mouth(52,39) | 2.48 (1.163) | 1.97 (1.088)
  Q7: Helping to Freshen Your Breath(n=50,33) | 2.28 (1.179) | 1.64 (1.025)
  Q8:Protecting Your Mouth From Drying Out(n=53,38) | 2.23 (1.137) | 1.84 (1.175)
  Q9: Providing Whole Mouth Comfort(n=53,38) | 2.38 (1.147) | 2.08 (1.148)
  Q10:Helping to Swallow Without Difficulty(n=51,36) | 2.37 (1.113) | 2.25 (1.339)
  Q11: Helping Mouth Feel 'Normal'(n=53,39) | 2.26 (1.163) | 2.08 (1.133)
  Q12:Having Long Lasting Dry Mouth Relief(n=51,38) | 2.27 (1.168) | 1.89 (1.110)
  Q13: Having a Long Lasting Lubricating Effect | 2.33 (1.227) | 1.85 (1.040)
  Q14: Having a Long Lasting moisturizing effect | 2.33 (1.160) | 1.92 (1.133)

15. Secondary Outcome: Mean Response to PPAQ1 at 5 Mins Post Treatment on Day 3
Description: Participants answered to the 3 questions in PPAQ1 as follows: Q1= Having a immediate dry mouth relief; Q2= Having a immediate lubricating effect; Q3= Having a immediate moisturizing effect. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 5 mins post treatment on Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 45
score on a scale
  Having a Immediate Dry Mouth Relief(n=53,45) | 3.55 (1.119) | 3.16 (1.397)
  Having a Immediate Lubricating Effect(n=53,44) | 3.47 (1.103) | 2.80 (1.440)
  Having a Immediate Moisturizing Effect(n=53,44) | 3.51 (1.067) | 2.89 (1.450)

16. Secondary Outcome: Mean Response to PPAQ2 at 30 Mins Post Treatment on Day 3
Description: Participants answered to the 11 questions in PPAQ2 as follows: Q1= Relieving the discomfort of dry mouth; Q2= Feeling comfortable in the mouth; Q3= Soothing your mouth; Q4= Allowing you to speak without difficulty; Q5= Effectively moistens your mouth; Q6= Effectively lubricates your mouth; Q7= Helping to freshen your breath; Q8= Protecting your mouth from drying out; Q9= Providing whole mouth comfort; Q10= Helping you to swallow without difficulty; Q11= Helping mouth feel normal. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 30 mins post treatment on Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort Of Dry Mouth(n=53,41) | 2.91 (1.043) | 2.29 (1.167)
  Q2:Feeling Comfortable in The Mouth(n=53,40) | 2.96 (1.055) | 2.35 (1.122)
  Q3:Soothing Your Mouth(n=53,40) | 2.91 (1.097) | 2.35 (1.272)
  Q4:Allowing to Speak Without Difficulty(n=46,36) | 3.11 (1.100) | 2.94 (1.286)
  Q5: Effectively Moistens Your Mouth(n= 53,42) | 2.92 (1.035) | 2.26 (1.270)
  Q6: Effectively Lubricates Your Mouth(53,40) | 2.85 (1.045) | 2.18 (1.259)
  Q7: Helping to Freshen Your Breath(n=53,33) | 2.94 (1.134) | 2.06 (1.197)
  Q8:Protecting Your Mouth From Drying Out(n=53,41) | 2.83 (1.122) | 2.02 (1.235)
  Q9: Providing Whole Mouth Comfort(n=53,42) | 2.87 (1.057) | 2.24 (1.246)
  Q10:Helping to Swallow Without Difficulty(n=49,41) | 3.00 (1.000) | 2.34 (1.257)
  Q11: Helping Mouth Feel 'Normal'(n=53,42) | 2.92 (1.053) | 2.24 (1.246)

17. Secondary Outcome: Mean Response to PPAQ3 at 60 Mins Post Treatment on Day 3
Description: Participants answered the 14 questions of PPAQ3 as follows: Q1= Relieving the discomfort of dry mouth; Q2= Feeling comfortable in the mouth; Q3= Soothing your mouth; Q4= Allowing you to speak without difficulty; Q5= Effectively moistens your mouth; Q6= Effectively lubricates your mouth; Q7= Helping to freshen your breath; Q8= Protecting your mouth from drying out; Q9= Providing whole mouth comfort; Q10= Helping you to swallow without difficulty; Q11= Helping mouth feel normal; Q12= Having a long lasting dry mouth relief; Q13= Having a long lasting lubricating effect; Q14= Having a long lasting moisturizing effect. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: 60 mins. post treatment on Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort of Dry Mouth(n=53,39) | 2.64 (1.058) | 2.10 (1.273)
  Q2:Feeling Comfortable in the Mouth(n=53,39) | 2.72 (1.133) | 2.21 (1.260)
  Q3:Soothing Your Mouth(n=53,39) | 2.66 (1.055) | 2.21 (1.281)
  Q4:Allowing to Speak Without Difficulty(n=46,35) | 2.89 (1.197) | 2.63 (1.285)
  Q5: Effectively Moistens Your Mouth(n= 53,40) | 2.60 (1.132) | 2.23 (1.230)
  Q6: Effectively Lubricates Your Mouth(53,39) | 2.60 (1.115) | 2.13 (1.361)
  Q7: Helping to Freshen Your Breath(n=52,34) | 2.75 (1.169) | 1.91 (1.190)
  Q8:Protecting Your Mouth From Drying Out(n=53,39) | 2.60 (1.132) | 1.92 (1.201)
  Q9: Providing Whole Mouth Comfort(n=53,40) | 2.75 (1.072) | 2.08 (1.269)
  Q10:Helping to Swallow Without Difficulty(n=49,37) | 2.65 (1.071) | 2.41 (1.235)
  Q11: Helping Mouth Feel 'Normal'(n=53,41) | 2.58 (1.046) | 2.20 (1.229)
  Q12:Having Long Lasting Dry Mouth Relief(n=53,39) | 2.55 (1.048) | 1.92 (1.326)
  Q13:Long Lasting Lubricating Effect(n=53,40) | 2.55 (1.048) | 2.00 (1.301)
  Q14:Long Lasting Moisturizing Effect(n=53,40) | 2.62 (1.096) | 1.98 (1.291)

18. Secondary Outcome: Mean Response to PPAQ3 at 120 Mins Post Treatment on Day 3
Description: as for outcome 14
Time Frame: 120 mins post treatment on Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort of Dry Mouth(n=53,39) | 2.60 (1.261) | 1.95 (1.297)
  Q2:Feeling Comfortable in the Mouth(n=53,41) | 2.57 (1.169) | 1.90 (1.114)
  Q3:Soothing Your Mouth(n=53,40) | 2.51 (1.234) | 1.93 (1.163)
  Q4:Allowing to Speak Without Difficulty(n=47,35) | 2.77 (1.127) | 2.51 (1.245)
  Q5: Effectively Moistens Your Mouth(n= 53,41) | 2.49 (1.203) | 1.93 (1.212)
  Q6: Effectively Lubricates Your Mouth(53,40) | 2.53 (1.219) | 1.95 (1.280)
  Q7: Helping to Freshen Your Breath(n=52,34) | 2.42 (1.242) | 1.79 (1.149)
  Q8:Protecting Your Mouth From Drying Out(n=53,38) | 2.45 (1.153) | 1.95 (1.184)
  Q9: Providing Whole Mouth Comfort(n=53,40) | 2.66 (1.208) | 1.90 (1.150)
  Q10:Helping to Swallow Without Difficulty(n=50,38) | 2.50 (1.233) | 2.16 (1.263)
  Q11: Helping Mouth Feel 'Normal'(n=53,39) | 2.55 (1.202) | 2.05 (1.213)
  Q12:Having Long Lasting Dry Mouth Relief(n=53,37) | 2.49 (1.234) | 1.89 (1.308)
  Q13:Long Lasting Lubricating Effect(n=53,39) | 2.43 (1.185) | 1.87 (1.260)
  Q14:Long Lasting Moisturizing Effect(n=53,41) | 2.45 (1.218) | 1.90 (1.281)

19. Secondary Outcome: Mean Response to PPAQ3 at 240 Mins Post Treatment on Day 3
Description: as for outcome 12
Time Frame: 240 mins post treatment on Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Q1:Relieving the Discomfort of Dry Mouth(n=52,39) | 2.37 (1.121) | 1.77 (1.180)
  Q2:Feeling Comfortable in the Mouth(n=52,40) | 2.42 (1.194) | 1.80 (1.043)
  Q3:Soothing Your Mouth(n=52,39) | 2.31 (1.130) | 1.77 (1.111)
  Q4:Allowing to Speak Without Difficulty(n=45,34) | 2.49 (1.121) | 2.26 (1.286)
  Q5: Effectively Moistens Your Mouth(n= 52,38) | 2.29 (1.143) | 1.76 (1.149)
  Q6: Effectively Lubricates Your Mouth(52,39) | 2.29 (1.160) | 1.74 (1.141)
  Q7: Helping to Freshen Your Breath(n=51,33) | 2.33 (1.178) | 1.76 (1.173)
  Q8:Protecting Your Mouth From Drying Out(n=52,39) | 2.25 (1.153) | 1.74 (1.117)
  Q9: Providing Whole Mouth Comfort(n=52,40) | 2.31 (1.164) | 1.75 (1.056)
  Q10:Helping to Swallow Without Difficulty(n=48,38) | 2.38 (1.123) | 1.92 (1.217)
  Q11: Helping Mouth Feel 'Normal'(n=52,38) | 2.33 (1.184) | 1.84 (1.103)
  Q12:Having Long Lasting Dry Mouth Relief(n=52,38) | 2.31 (1.164) | 1.71 (1.206)
  Q13:Long Lasting Lubricating Effect(n=52,39) | 2.23 (1.165) | 1.72 (1.169)
  Q14:Long Lasting Moisturizing Effect(n=52,39) | 2.23 (1.148) | 1.77 (1.158)

20. Secondary Outcome: Mean Response to PPAQ4 Prior to Treatment on Day 3
Description: Participants answered to the 9 questions in PPAQ4. Q1= Providing relief all night; Q2= Reducing the number of times you wake up from dry mouth; Q3= Feeling less parched when you wake up; Q4= Having a long lasting dry mouth relief; Q5= Having a long lasting lubricating effect; Q6= Having a long lasting moisturizing effect; Q7= Having an overall dry mouth relief; Q8= Having an overall lubrication effect; Q9= Having an overall moisturizing effect. These questions were rated on scale as follows: N/A = Not Applicable; 1 = poor; 2 = fair; 3 = good; 4 = very good; 5 = excellent. Scale score was averaged to calculate the response.
Time Frame: Prior to treatment on Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Providing Relief All Night(n=51,34) | 2.57 (1.100) | 2.18 (1.336)
  Reducing Number of Wake Up from Dry Mouth(n=47,33) | 2.81 (1.173) | 2.18 (1.334)
  Feeling Less Parched When You Wake Up(n=50,36) | 2.52 (1.129) | 2.11 (1.214)
  Having a Long Lasting Dry Mouth Relief(n=53,36) | 2.43 (1.047) | 1.86 (1.125)
  Having a Long Lasting Lubricating Effect(n=53,36) | 2.51 (1.067) | 2.00 (1.219)
  Having a Long Lasting Moisturizing Effect(n=53,36) | 2.47 (1.012) | 1.86 (1.150)
  Having an Overall Dry Mouth Relief(n=53,37) | 2.45 (1.048) | 1.95 (1.177)
  Having an Overall Lubrication Effect(n=53,36) | 2.47 (1.049) | 2.03 (1.183)
  Having an Overall Moisturizing Effect(n=53,37) | 2.45 (1.084) | 2.03 (1.166)

21. Secondary Outcome: Mean Response to Subjective Assessment of Patient's Quality of Life (SAoP QoL1) Prior to Treatment on Day 1
Description: Participants answered to the 6 questions in SAoP QoL as follows: Q1= Does your dry mouth cause discomfort?; Q2= Does your dry mouth make it uncomfortable to speak?; Q3= Does your dry mouth interrupt your sleep?; Q4= Does your dry mouth affect your social interactions?; Q5= Does your dry mouth cause you to avoid certain foods?; Q6= Does your dry mouth interfere with your daily activities? These questions were rated on a scale as follows: 0 = not at all; 1 = a little; 2 = somewhat; 3 = quite a bit; 4 = very much. Scale score was averaged to calculate the response.
Time Frame: Prior to treatment on Day 1
Population: Analysis for this outcome was conducted on ITT population which included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Does Your Dry Mouth Cause Discomfort? | 2.51 (1.310) | 2.74 (1.073)
  Does Your Dry Mouth Make Uncomfortable To Speak? | 2.13 (1.256) | 2.06 (1.111)
  Does Your Dry Mouth Interrupt Your Sleep? | 2.08 (1.253) | 2.13 (1.454)
  Does Your Dry Mouth Affect Your Social Interaction | 1.58 (1.247) | 1.51 (1.349)
  Does Your Dry Mouth Cause To Avoid Certain Foods? | 1.87 (1.532) | 1.94 (1.451)
  Does Dry Mouth Interfere Your Daily Activities? | 1.42 (1.322) | 1.36 (1.326)

22. Secondary Outcome: Mean Response to SAoP QoL 2 Prior to Treatment on Day 8
Description: Participants answered to the 6 questions in SAoP QoL 2 as follows: Q1= Looking back over the last 7 days, has your dry mouth caused discomfort?; Q2= Looking back over the last 7 days, has your dry mouth made it uncomfortable to speak?; Q3= Looking back over the last 7 days, has your dry mouth interrupted your sleep?; Q4= Looking back over the last 7 days, has your dry mouth affected your social interactions?; Q5= Looking back over the last 7 days, has your dry mouth caused you to avoid certain foods?; Q6= Looking back over the last 7 days, has your dry mouth interfered with your daily activities? These questions were rated on scale as follows: 0 = not at all; 1 = a little; 2 = somewhat; 3 = quite a bit; 4 = very much. Scale score was averaged to calculate the response.
Time Frame: prior to treatment on Day 8
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Has Your Dry Mouth Cause Discomfort? | 1.58 (1.216) | 2.15 (1.215)
  Has Your Dry Mouth Make Uncomfortable To Speak? | 1.00 (1.127) | 1.32 (1.144)
  Has Your Dry Mouth Interrupt Your Sleep? | 1.15 (1.215) | 1.66 (1.493)
  Has Your Dry Mouth Affect Social Interactions? | 0.70 (1.030) | 1.02 (1.242)
  Has Your Dry Mouth Cause To Avoid Certain Foods? | 1.11 (1.368) | 1.49 (1.333)
  Has Your Mouth Interfere Daily Activities? | 0.83 (1.033) | 0.87 (1.227)

23. Secondary Outcome: Number of Participants With Response to Dry Mouth Inventory Quality of Life (DMI QoL) Question (Q) Numbers 1 to 15 on Day 1
Description: Number of Participants were reported who answered following questions, Q1:Thinking back during last week, how often has your dry mouth been a problem? Having a dry mouth affects people in different ways. Please tell us how much you agree or disagree whether your dry mouth has affected you in these ways in last week Q2:Rawness or soreness? Q3:Uncomfortable? Q4:Bad taste? Q5:Loss of taste? Q6:Lips sticking to teeth? Q7:Tongue sticking to roof of mouth? Q8:Throat dry? Q9:No moisture? Q10:Mouth feels tight? Dry mouth stops some people doing things. How much do you agree or disagree that it has been difficult for you to do following things in last week? Q11:Eating dry foods? Q12:Eating sticky foods? Q13:Eating hard or scratchy foods such as crisps, biscuits or nuts?, How much do you recognize yourself in following statements, based on the last week? Q14:Swallowing has been difficult for me this last week? Q15:Drinking so much means that I go to the toilet more than other people?
Time Frame: Prior to treatment on Day 1
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q1:Never in the last week | 3 | 2
  Q1: A few days | 10 | 5
  Q1:Most days | 9 | 6
  Q1: Every day | 13 | 11
  Q1: Several times every day | 8 | 11
  Q1: All of the time | 10 | 12
  Q2: Strongly disagree | 8 | 8
  Q2: Disagree | 12 | 12
  Q2: Disagree a little | 5 | 6
  Q2: Agree a little | 13 | 6
  Q2: Agree | 14 | 10
  Q2: Strongly Agree | 1 | 5
  Q3: Strongly disagree | 3 | 2
  Q3: Disagree | 2 | 0
  Q3: Disagree a little | 2 | 2
  Q3: Agree a little | 7 | 9
  Q3: Agree | 26 | 23
  Q3: Strongly agree | 13 | 11
  Q4: Strongly disagree | 2 | 3
  Q4: Disagree | 5 | 6
  Q4: Disagree a little | 5 | 4
  Q4: Agree a little | 15 | 10
  Q4: Agree | 16 | 15
  Q4: Strongly agree | 10 | 9
  Q5: Strongly disagree | 7 | 8
  Q5: Disagree | 10 | 10
  Q5: Disagree a little | 4 | 4
  Q5: Agree a little | 14 | 11
  Q5:Agree | 11 | 10
  Q5: Strongly Agree | 7 | 4
  Q6: Strongly disagree | 5 | 4
  Q6: Disagree | 3 | 3
  Q6:Disagree a little | 4 | 7
  Q6: Agree a little | 18 | 9
  Q6: Agree | 16 | 15
  Q6: Strongly agree | 7 | 9
  Q7: Strongly disagree | 5 | 5
  Q7: Disagree | 5 | 3
  Q7: Disagree a little | 6 | 4
  Q7: Agree a little | 17 | 10
  Q7: Agree | 14 | 15
  Q7: Strongly agree | 6 | 10
  Q8: Strongly disagree | 0 | 1
  Q8: Disagree | 2 | 1
  Q8: Disagree a little | 2 | 0
  Q8: Agree a little | 12 | 9
  Q8: Agree | 21 | 20
  Q8: Strongly agree | 16 | 16
  Q9: Strongly disagree | 1 | 0
  Q9: Disagree | 1 | 2
  Q9: Disagree a little | 2 | 0
  Q9: Agree a little | 9 | 10
  Q9: Agree | 22 | 20
  Q9: Strongly agree | 18 | 15
  Q10: Strongly disagree | 3 | 2
  Q10: Disagree | 9 | 6
  Q10: Disagree a little | 5 | 3
  Q10: Agree a little | 10 | 12
  Q10: Agree | 15 | 16
  Q10: Strongly agree | 11 | 8
  Q11: Strongly disagree | 2 | 3
  Q11: Disagree | 5 | 6
  Q11: Disagree a little | 1 | 4
  Q11: Agree a little | 18 | 10
  Q11: Agree | 13 | 9
  Q11: Strongly agree | 14 | 15
  Q12: Strongly diaagree | 3 | 3
  Q12: Disagree | 7 | 6
  Q12: Disagree a little | 3 | 3
  Q12: Agree a little | 17 | 11
  Q12: Agree | 13 | 16
  Q12: Strongly agree | 10 | 8
  Q13: Strongly disagree | 2 | 3
  Q13: Disagree | 3 | 4
  Q13: Disagree a little | 7 | 2
  Q13: Agree a little | 14 | 10
  Q13: Agree | 11 | 13
  Q13: Strongly agree | 16 | 15
  Q14: Strongly disagree | 3 | 5
  Q14: Disagree | 7 | 6
  Q14: Disagree a little | 4 | 4
  Q14: Agree a little | 14 | 13
  Q14: Agree | 18 | 15
  Q14: Strongly agree | 7 | 4
  Q15: Strongly disagree | 2 | 0
  Q15: Disagree | 5 | 4
  Q15: Disagree a little | 1 | 6
  Q15: Agree a little | 9 | 6
  Q15: Agree | 8 | 13
  Q15: Strongly agree | 28 | 18

24. Secondary Outcome: Number of Participants With Responses to DMI QoL Question(Q) Numbers 16 to 27 on Day 1
Description: Number of Participants were reported who answered following questions, how often during last week has a dry mouth affected these aspects of your life? Q16:My dry mouth interrupts my sleep; Q17:My dry mouth makes it difficult for me to speak; Q18:My dry mouth interferes with me being intimate with those close to me; Q19:My dry mouth means it takes me longer to eat meals, Having a dry mouth can affect people's moods & emotions. Please tell us how much you agree or disagree that your dry mouth has given you these moods over last week; Q20:Irritable; Q21:Worried; Q22:Frustrated; Q23:Always on my mind; Q24:It gets me down, How much do you agree or disagree that your dry mouth has affected your time with other people over the last week?; Q25:Drinking or going to the toilet interrupts my conversations; Q26:I have difficulty using the telephone; Q27:I feel different because of the things I have to do to look after my mouth.
Time Frame: Prior to treatment on Day 1
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q16: Never | 11 | 7
  Q16: A few days | 14 | 19
  Q16: Most days | 9 | 6
  Q16: Every day | 6 | 4
  Q16: A few times every day | 2 | 5
  Q16: Many times every day | 11 | 6
  Q17: Never | 16 | 13
  Q17: A few days | 7 | 14
  Q17: Most days | 9 | 8
  Q17: Every day | 6 | 3
  Q17: A few times every day | 10 | 6
  Q17: Many times every day | 5 | 3
  Q18: Never | 22 | 19
  Q18: A few days | 12 | 7
  Q18: Most days | 5 | 9
  Q18: Every day | 4 | 3
  Q18: A few times every day | 4 | 5
  Q18: Many times every day | 6 | 4
  Q19: Never | 21 | 13
  Q19: A few days | 8 | 12
  Q19: Most days | 6 | 6
  Q19: Every day | 6 | 6
  Q19: A few times every day | 2 | 6
  Q19: Many times every day | 10 | 4
  Q20: Strongly disagree | 10 | 6
  Q20: Disagree | 8 | 9
  Q20: Disagree a little | 4 | 6
  Q20: Agree a little | 18 | 16
  Q20: Agree | 8 | 7
  Q20: Strongly agree | 5 | 3
  Q21: Strongly disagree | 8 | 8
  Q21: Disagree | 9 | 14
  Q21: Disagree a little | 4 | 6
  Q21: Agree a little | 16 | 6
  Q21: Agree | 11 | 7
  Q21: Strongly agree | 5 | 6
  Q22: Strongly disagree | 8 | 5
  Q22: Disagree | 8 | 10
  Q22: Disagree a little | 6 | 1
  Q22: Agree a little | 8 | 11
  Q22: Agree | 16 | 15
  Q22: Strongly agree | 7 | 5
  Q23: Strongly disagree | 7 | 5
  Q23: Disagree | 7 | 9
  Q23: Disagree a little | 8 | 4
  Q23: Agree a little | 10 | 11
  Q23: Agree | 12 | 12
  Q23: Strongly agree | 9 | 6
  Q24: Strongly disagree | 7 | 8
  Q24: Disagree | 13 | 9
  Q24: Disagree a little | 9 | 7
  Q24: Agree a little | 13 | 9
  Q24: Agree | 6 | 7
  Q24: Strongly agree | 5 | 7
  Q25: Strongly disagree | 5 | 6
  Q25: Disagree | 10 | 5
  Q25: Disagree a little | 6 | 6
  Q25: Agree a little | 12 | 12
  Q25: Agree | 8 | 12
  Q25: Strongly agree | 12 | 6
  Q26: Strongly disagree | 9 | 7
  Q26: Disagree | 9 | 16
  Q26:Disagree a little | 9 | 7
  Q26: Agree a little | 20 | 11
  Q26: Agree | 3 | 4
  Q26: Strongly agree | 3 | 2
  Q27: Strongly disagree | 6 | 9
  Q27: Disagree | 11 | 7
  Q27: Disagree a little | 7 | 7
  Q27: Agree a little | 13 | 12
  Q27: Agree | 11 | 8
  Q27: Strongly agree | 5 | 4

25. Secondary Outcome: Number of Participants With Response to DMI QoL Question (Q) Number 28 to 39 on Day 1
Description: Number of participants were reported who answered following questions, these questions were about how participants had coped with their dry mouth over the last week with respect to agree or disagree with each of the following questions. Q28:I have to drink a lot of water; Q29:I need to carry water with me everywhere I go; Q30:I worry about where I can go to the toilet; Q31:I have to drink something with food; Q32:I have to clean my teeth more than most people; Q33:I choose moist foods when I can; Q34:I need sauces to help me eat; Q35:I avoid certain foods or drinks, and There are other things that help some people with dry mouth. Please tell us how often over the last week, that you have done these things. Q36:I have chewed gum; Q37:I have chewed my food for longer; Q38:I have sucked sweets or mints or pastilles; Q39:I have breathed through my nose rather than my mouth.
Time Frame: Prior to treatment on Day 1
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q28: Strongly disagree | 2 | 0
  Q28: Disagree | 1 | 1
  Q28: Disagree a little | 0 | 1
  Q28: Agree a little | 4 | 5
  Q28: Agree | 14 | 13
  Q28: Strongly agree | 32 | 27
  Q29: Strongly disagree | 4 | 1
  Q29: Disagree | 5 | 0
  Q29: Disagree a little | 0 | 5
  Q29: Agree a little | 6 | 8
  Q29: Agree | 16 | 14
  Q29: Strongly agree | 22 | 19
  Q30: Strongly disagree | 4 | 2
  Q30: Disagree | 3 | 5
  Q30: Disagree a little | 3 | 3
  Q30: Agree a little | 12 | 13
  Q30: Agree | 10 | 11
  Q30: Strongly agree | 21 | 13
  Q31: Strongly disagree | 3 | 2
  Q31: Disagree | 0 | 2
  Q31: Disagree a little | 2 | 0
  Q31: Agree a little | 5 | 5
  Q31: Agree | 14 | 9
  Q31: Strongly agree | 29 | 29
  Q32: Strongly disagree | 4 | 2
  Q32: Disagree | 6 | 5
  Q32: Disagree a little | 2 | 3
  Q32: Agree a little | 15 | 12
  Q32: Agree | 14 | 14
  Q32: Strongly agree | 12 | 11
  Q33: Strongly disagree | 2 | 1
  Q33: Disagree | 6 | 3
  Q33: Disagree a little | 6 | 4
  Q33: Agree a little | 12 | 7
  Q33: Agree | 15 | 20
  Q33: Strongly agree | 12 | 12
  Q34: Strongly disagree | 6 | 2
  Q34: Disagree | 12 | 11
  Q34: Disagree a little | 5 | 6
  Q34: Agree a little | 11 | 9
  Q34: Agree | 10 | 11
  Q34: Strongly agree | 9 | 8
  Q35: Strongly disagree | 6 | 2
  Q35: Disagree | 11 | 7
  Q35: Disagree a little | 4 | 5
  Q35: Agree a little | 6 | 8
  Q35: Agree | 14 | 12
  Q35: Strongly agree | 12 | 13
  Q36: Never in the last week | 20 | 17
  Q36: One or two days | 5 | 7
  Q36: Most days | 10 | 7
  Q36: Every day | 3 | 1
  Q36: A few times every day | 6 | 5
  Q36: Many times every day | 9 | 10
  Q37: Never in the last week | 7 | 8
  Q37: One or two days | 8 | 9
  Q37: Most days | 9 | 7
  Q37: Every day | 10 | 10
  Q37: A few times every day | 6 | 5
  Q37: Many times every day | 13 | 8
  Q38: Never in the last week | 13 | 12
  Q38: One or two days | 8 | 11
  Q38: Most days | 8 | 5
  Q38: Every day | 8 | 4
  Q38: A few times every day | 10 | 4
  Q38: Many times every day | 6 | 11
  Q39: Never in the last week | 10 | 11
  Q39: One or two days | 6 | 3
  Q39: Most days | 10 | 7
  Q39: Every day | 8 | 9
  Q39: A few times every day | 6 | 3
  Q39: Many times every day | 13 | 14

26. Secondary Outcome: Number of Participants With Response to DMI QoL Question (Q) Number 40 to 46 and QM1-QM8 on Day 1
Description: Number Participants were reported who answered following questions with respect to how much they agree or disagree with following statements over the last week & how much they agreed that symptoms were manageable (M). Q40:It's a big issue for me; Q41:My dry mouth makes me feel different to other people; Q42:My mouth is deteriorating, Dry mouth can also affect your quality of life; Q43:Dry mouth is part of my life nowadays; Q44:Dry mouth is a quality of life issue; Q45:My dry mouth stops me enjoying things; Q46:How would you rate your oral health overall?, and Think back over last week about things you have done to relieve your symptoms. How much do you agree or disagree that those things have made following symptoms more manageable? M1: Uncomfortable; M2: Bad taste; M3:Loss of Taste; M4: Lips sticking to roof of mouth; M5: Tongue sticking to roof of mouth; M6: Throat dry; M7: No moisture M8:Devoid of any wetness M9:Mouth feels tight ?
Time Frame: Prior to treatment on Day 1
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q40: Strongly Disagree | 3 | 3
  Q40: Disagree | 6 | 6
  Q40: Disagree a little | 2 | 4
  Q40: Agree a little | 13 | 11
  Q40: Agree | 17 | 16
  Q40: Strongly agree | 12 | 7
  Q41: Strongly disagree | 5 | 7
  Q41: Disagree | 12 | 11
  Q41: Disagree a little | 6 | 7
  Q41: Agree a little | 15 | 4
  Q41: Agree | 6 | 12
  Q41: Strongly agree | 9 | 6
  Q42: Strongly disagree | 6 | 4
  Q42: Disagree | 12 | 7
  Q42: Disagree a little | 3 | 6
  Q42: Agree a little | 15 | 11
  Q42: Agree | 6 | 11
  Q42: Strongly agree | 11 | 8
  Q43: Strongly disagree | 2 | 2
  Q43: Disagree | 2 | 1
  Q43: Disagree a little | 3 | 0
  Q43: Agree a little | 10 | 10
  Q43: Agree | 16 | 21
  Q43: Strongly agree | 20 | 13
  Q44: Strongly disagree | 2 | 2
  Q44: Disagree | 8 | 2
  Q44: Disagree a little | 4 | 6
  Q44: Agree a little | 12 | 14
  Q44: Agree | 13 | 14
  Q44: Strongly agree | 14 | 9
  Q45: Strongly disagree | 6 | 4
  Q45: Disagree | 12 | 10
  Q45: Disagree a little | 7 | 8
  Q45: Agree a little | 14 | 9
  Q45: Agree | 6 | 10
  Q45: Strongly agree | 8 | 6
  Q46: Excellent | 5 | 3
  Q46: Very Good | 12 | 10
  Q46: Good | 20 | 14
  Q46: Fair | 13 | 15
  Q46: Poor | 3 | 5
  QM1: Strongly disagree | 2 | 2
  QM1: Disagree | 9 | 1
  QM1: Disagree a little | 5 | 4
  QM1: Agree a little | 17 | 12
  QM1: Agree | 15 | 17
  QM1: Strongly agree | 5 | 11
  QM2: Strongly disagree | 4 | 4
  QM2: Disagree | 11 | 4
  QM2: Disagree a little | 8 | 3
  QM2: Agree a little | 13 | 13
  QM2: Agree | 11 | 15
  QM2: Strongly agree | 6 | 8
  QM3: Strongly disagree | 5 | 6
  QM3: Disagree | 17 | 5
  QM3: Disagree a little | 8 | 12
  QM3: Agree a little | 12 | 12
  QM3: Agree | 9 | 11
  QM3: Strongly agree | 2 | 1
  QM4: Strongly disagree | 5 | 3
  QM4: Disagree | 10 | 3
  QM4: Disagree a little | 6 | 5
  QM4: Agree a little | 17 | 11
  QM4: Agree | 11 | 17
  QM4: Strongly agree | 4 | 8
  QM5: Strongly disagree | 6 | 3
  QM5: Disagree | 9 | 3
  QM5: Disagree a little | 6 | 4
  QM5: Agree a little | 16 | 11
  QM5: Agree | 13 | 16
  QM5: Strongly agree | 3 | 10
  QM6: Strongly disagree | 1 | 1
  QM6: Disagree | 7 | 1
  QM6: Disagree a little | 2 | 3
  QM6: Agree a little | 18 | 9
  QM6: Agree | 17 | 17
  QM6: Strongly agree | 8 | 16
  QM7: Strongly disagree | 3 | 0
  QM7: Disagree | 7 | 3
  QM7: Disagree a little | 2 | 4
  QM7: Agree a little | 15 | 7
  QM7: Agree | 16 | 17
  QM7: Strongly agree | 10 | 16
  QM8: Strongly disagree | 3 | 2
  QM8: Disagree | 7 | 4
  QM8: Disagree a little | 5 | 4
  QM8: Agree a little | 16 | 7
  QM8: Agree | 15 | 22
  QM8: Strongly agree | 7 | 8
  QM9: Strongly disagree | 6 | 4
  QM9: Disagree | 13 | 3
  QM9: Disagree a little | 6 | 4
  QM9: Agree a little | 12 | 11
  QM9: Agree | 10 | 18
  QM9: Strongly agree | 6 | 7

27. Secondary Outcome: Number of Participants With Responses to DMI QoL Question(Q) Numbers 1 to 15 on Day 8
Description: Number of participants were reported who answered following questions, Q1:Thinking back during last week, how often has your dry mouth been a problem?; Having a dry mouth affects people in different ways. Please tell us how much you agree or disagree whether your dry mouth has affected you in these ways in last week Q2:Rawness or soreness? Q3:Uncomfortable? Q4:Bad taste? Q5:Loss of taste? Q6:Lips sticking to teeth? Q7:Tongue sticking to roof of mouth? Q8:Throat dry? Q9:No moisture? Q10:Mouth feels tight? Dry mouth stops some people doing things. How much do you agree or disagree that it has been difficult for you to do following things in last week? Q11:Eating dry foods? Q12:Eating sticky foods? Q13:Eating hard or scratchy foods such as crisps, biscuits or nuts?, and How much do you recognize yourself in following statements, based on last week? Q14:Swallowing has been difficult for me this last week? Q15:Drinking so much means that I go to the toilet more than other people?
Time Frame: Prior to treatment on Day 8
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q1: Never in the last week | 8 | 2
  Q1: A few days | 20 | 8
  Q1: Most days | 7 | 14
  Q1: Every day | 7 | 10
  Q1: Several times every day | 3 | 8
  Q1: All of the time | 8 | 5
  Q2: Strongly disagree | 14 | 12
  Q2: Disagree | 11 | 11
  Q2: Disagree a little | 4 | 6
  Q2: Agree a little | 13 | 7
  Q2: Agree | 9 | 9
  Q2: Strongly agree | 2 | 2
  Q3: Strongly disagree | 6 | 5
  Q3: Disagree | 6 | 2
  Q3: Disagree a little | 8 | 2
  Q3: Agree a little | 12 | 9
  Q3: Agree | 13 | 21
  Q3: Strongly agree | 8 | 8
  Q4: Strongly disagree | 6 | 7
  Q4: Disagree | 6 | 7
  Q4: Disagree a little | 7 | 3
  Q4: Agree a little | 19 | 11
  Q4: Agree | 12 | 12
  Q4: Strongly agree | 3 | 7
  Q5: Strongly disagree | 13 | 11
  Q5: Disagree | 13 | 12
  Q5: Disagree a little | 6 | 7
  Q5: Agree a little | 14 | 6
  Q5: Agree | 5 | 8
  Q5: Strongly agree | 2 | 3
  Q6: Strongly disagree | 9 | 5
  Q6: Disagree | 7 | 3
  Q6: Disagree a little | 7 | 8
  Q6: Agree a little | 14 | 9
  Q6: Agree | 12 | 15
  Q6: Strongly agree | 4 | 7
  Q7: Strongly disagree | 11 | 3
  Q7: Disagree | 9 | 5
  Q7: Disagree a little | 9 | 10
  Q7: Agree a little | 14 | 8
  Q7: Agree | 9 | 16
  Q7: Strongly agree | 1 | 5
  Q8: Strongly disagree | 3 | 4
  Q8: Disagree | 3 | 1
  Q8: Disagree a little | 4 | 2
  Q8: Agree a little | 17 | 9
  Q8: Agree | 16 | 18
  Q8: Strongly agree | 10 | 13
  Q9: Strongly disagree | 4 | 3
  Q9: Disagree | 4 | 4
  Q9: Disagree a little | 5 | 0
  Q9: Agree a little | 14 | 9
  Q9: Agree | 14 | 21
  Q9: Strongly agree | 12 | 10
  Q10: Strongly disagree | 8 | 4
  Q10: Disagree | 8 | 5
  Q10: Disagree a little | 7 | 3
  Q10: Agree a little | 12 | 14
  Q10: Agree | 12 | 15
  Q10: Strongly agree | 6 | 6
  Q11: Strongly disagree | 6 | 4
  Q11: Disagree | 10 | 8
  Q11: Disagree a little | 7 | 3
  Q11: Agree a little | 13 | 10
  Q11: Agree | 11 | 16
  Q11: Strongly agree | 6 | 6
  Q12: Strongly disagree | 7 | 2
  Q12: Disagree | 11 | 11
  Q12: Disagree a little | 10 | 5
  Q12: Agree a little | 14 | 11
  Q12: Agree | 8 | 13
  Q12: Strongly agree | 3 | 5
  Q13: Strongly disagree | 6 | 4
  Q13: Disagree | 11 | 9
  Q13: Disagree a little | 11 | 1
  Q13: Agree a little | 15 | 10
  Q13: Agree | 5 | 14
  Q13: Strongly agree | 5 | 9
  Q14: Strongly disagree | 6 | 5
  Q14: Disagree | 14 | 13
  Q14: Disagree a little | 11 | 6
  Q14: Agree a little | 12 | 12
  Q14: Agree | 9 | 8
  Q14: Strongly agree | 1 | 3
  Q15: Strongly disagree | 5 | 5
  Q15: Disagree | 7 | 5
  Q15: Disagree a little | 6 | 0
  Q15: Agree a little | 13 | 7
  Q15: Agree | 12 | 16
  Q15: Strongly agree | 10 | 14

28. Secondary Outcome: Number of Participants With Responses to DMI QoL Question(Q) Numbers 16 to 27 on Day 8
Description: Number of participants were reported who answered following questions, how often during last week has a dry mouth affected these aspects of your life? Q16:My dry mouth interrupts my sleep; Q17:My dry mouth makes it difficult for me to speak; Q18:My dry mouth interferes with me being intimate with those close to me; Q19:My dry mouth means it takes me longer to eat meals, Having a dry mouth can affect people's moods and emotions. Please tell us how much you agree or disagree that your dry mouth has given you these moods over the last week Q20:Irritable; Q21:Worried; Q22:Frustrated; Q23:Always on my mind; Q24:It gets me down, and How much do you agree or disagree that your dry mouth has affected your time with other people over last week? Q25:Drinking or going to the toilet interrupts my conversations; Q26:I have difficulty using the telephone Q27:I feel different because of the things I have to do to look after my mouth.
Time Frame: Prior to treatment on Day 8
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q16: Never | 16 | 15
  Q16: A few days | 21 | 9
  Q16: Most days | 8 | 6
  Q16: Every day | 3 | 7
  Q16: A few times every day | 2 | 6
  Q16: Many times every day | 3 | 4
  Q17: Never | 20 | 12
  Q17: A few days | 20 | 20
  Q17: Most days | 8 | 3
  Q17: Every day | 0 | 3
  Q17: A few times every day | 3 | 8
  Q17: Many times every day | 2 | 1
  Q18: Never | 33 | 19
  Q18: A few days | 12 | 15
  Q18: Most days | 2 | 5
  Q18: Every day | 3 | 2
  Q18: A few times every day | 1 | 3
  Q18: Many times every day | 2 | 3
  Q19: Never | 23 | 15
  Q19: A few days | 13 | 8
  Q19: Most days | 7 | 11
  Q19: Every day | 7 | 8
  Q19: A few times every day | 2 | 2
  Q19: Many times every day | 1 | 3
  Q20: Strongly disagree | 14 | 13
  Q20: Disagree | 17 | 13
  Q20: Disagree a little | 3 | 5
  Q20: Agree a little | 12 | 7
  Q20: Agree | 7 | 7
  Q20: Strongly agree | 0 | 2
  Q21: Strongly disagree | 13 | 11
  Q21: Disagree | 18 | 10
  Q21: Disagree a little | 1 | 8
  Q21: Agree a little | 14 | 7
  Q21: Agree | 6 | 8
  Q21: Strongly agree | 1 | 3
  Q22: Strongly disagree | 11 | 10
  Q22: Disagree | 14 | 10
  Q22: Disagree a little | 3 | 5
  Q22: Agree a little | 17 | 7
  Q22: Agree | 7 | 12
  Q22: Strongly agree | 1 | 3
  Q23: Strongly disagree | 11 | 9
  Q23: Disagree | 14 | 8
  Q23: Disagree a little | 4 | 4
  Q23: Agree a little | 13 | 10
  Q23: Agree | 7 | 11
  Q23: Strongly agree | 4 | 5
  Q24: Strongly disagree | 13 | 12
  Q24: Disagree | 15 | 9
  Q24: Disagree a little | 4 | 8
  Q24: Agree a little | 14 | 8
  Q24: Agree | 4 | 8
  Q24: Strongly agree | 3 | 2
  Q25: Strongly disagree | 10 | 7
  Q25: Disagree | 9 | 8
  Q25: Disagree a little | 9 | 3
  Q25: Agree a little | 12 | 11
  Q25: Agree | 9 | 13
  Q25: Strongly agree | 4 | 5
  Q26: Strongly disagree | 15 | 12
  Q26: Disagree | 15 | 10
  Q26: Disagree a little | 5 | 10
  Q26: Agree a little | 16 | 11
  Q26: Agree | 2 | 2
  Q26: Strongly agree | 0 | 2
  Q27: Strongly disagree | 12 | 12
  Q27: Disagree | 14 | 9
  Q27: Disagree a little | 2 | 2
  Q27: Agree a little | 17 | 10
  Q27: Agree | 7 | 8
  Q27: Strongly agree | 1 | 6

29. Secondary Outcome: Number of Participants With Response to DMI QoL Question(Q) Numbers 28 to 39 on Day 8
Description: Number of participants were reported who answered following questions, these questions are about how you have coped with your dry mouth over last week. Please tell us whether you agree or disagree with each of the statements. Q28:I have to drink a lot of water; Q29:I need to carry water with me everywhere I go; Q30:I worry about where I can go to toilet; Q31:I have to drink something with food; Q32:I have to clean my teeth more than most people; Q33:I choose moist foods when I can; Q34:I need sauces to help me eat; Q35:I avoid certain foods or drinks, There are other things that help some people with dry mouth. Please tell us how often over last week, that you have done these things. Q36:I have chewed gum; Q37:I have chewed my food for longer; Q38:I have sucked sweets or mints or pastilles; Q39:I have breathed through my nose rather than my mouth.
Time Frame: Prior to treatment on Day 8
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q28: Strongly disagree | 2 | 2
  Q28: Disagree | 0 | 1
  Q28: Disagree a little | 5 | 3
  Q28: Agree a little | 15 | 3
  Q28: Agree | 11 | 14
  Q28: Strongly agree | 20 | 24
  Q29: Strongly disagree | 4 | 1
  Q29: Disagree | 9 | 2
  Q29: Disagree a little | 6 | 3
  Q29: Agree a little | 12 | 10
  Q29: Agree | 12 | 12
  Q29: Strongly agree | 10 | 19
  Q30: Strongly disagree | 7 | 3
  Q30: Disagree | 5 | 7
  Q30: Disagree a little | 4 | 4
  Q30: Agree a little | 20 | 10
  Q30: Agree | 10 | 13
  Q30: Strongly agree | 7 | 10
  Q31: Strongly disagree | 6 | 2
  Q31: Disagree | 1 | 2
  Q31: Disagree a little | 1 | 2
  Q31: Agree a little | 9 | 6
  Q31: Agree | 16 | 14
  Q31: Strongly agree | 20 | 21
  Q32: Strongly disagree | 6 | 3
  Q32: Disagree | 6 | 4
  Q32: Disagree a little | 8 | 7
  Q32: Agree a little | 12 | 12
  Q32: Agree | 12 | 12
  Q32: Strongly agree | 9 | 9
  Q33: Strongly disagree | 6 | 1
  Q33: Disagree | 6 | 5
  Q33: Disagree a little | 6 | 4
  Q33: Agree a little | 13 | 10
  Q33: Agree | 15 | 17
  Q33: Strongly agree | 7 | 10
  Q34: Strongly disagree | 10 | 2
  Q34: Disagree | 8 | 10
  Q34: Disagree a little | 10 | 7
  Q34: Agree a little | 15 | 7
  Q34: Agree | 7 | 11
  Q34: Strongly agree | 3 | 10
  Q35: Strongly disagree | 10 | 4
  Q35: Disagree | 9 | 8
  Q35: Disagree a little | 7 | 4
  Q35: Agree a little | 13 | 5
  Q35: Agree | 6 | 10
  Q35: Strongly agree | 8 | 16
  Q36: Never in the last week | 38 | 22
  Q36: One or two days | 5 | 4
  Q36: Most days | 4 | 7
  Q36: Every day | 2 | 2
  Q36: A few times every day | 1 | 5
  Q36: Many times every day | 3 | 7
  Q37: Never in the last week | 20 | 11
  Q37: One or two days | 10 | 9
  Q37: Most days | 9 | 8
  Q37: Every day | 9 | 9
  Q37: A few times every day | 2 | 2
  Q37: Many times every day | 3 | 8
  Q38: Never in the last week | 31 | 19
  Q38: One or two days | 10 | 3
  Q38: Most days | 3 | 7
  Q38: Every day | 7 | 6
  Q38: A few times every day | 0 | 2
  Q38: Many times every day | 2 | 10
  Q39: Never in the last week | 23 | 7
  Q39: One or two days | 6 | 11
  Q39: Most days | 7 | 6
  Q39: Every day | 8 | 6
  Q39: A few times every day | 2 | 2
  Q39: Many times every day | 7 | 15

30. Secondary Outcome: Number of Participants With Response to DMI QoL Question (Q) Number 40 to 46 and QM1- QM9 on Day 8
Description: Number Participants were reported who answered following questions with respect to how much they agree or disagree with following statements over the last week & how much they agreed that symptoms were manageable (M). Q40:It's a big issue for me; Q41:My dry mouth makes me feel different to other people; Q42:My mouth is deteriorating, Dry mouth can also affect your quality of life. Q43:Dry mouth is part of my life nowadays; Q44:Dry mouth is a quality of life issue; Q45:My dry mouth stops me enjoying things; Q46:How would you rate your oral health overall?, and Think back over last week about things you have done to relieve your symptoms. How much do you agree or disagree that those things have made following symptoms more manageable? M1:Uncomfortable; M2:Bad taste; M3:Loss of Taste; M4:Lips sticking to roof of mouth; M5:Tongue sticking to roof of mouth; M6: Throat dry; M7:No moisture; M8:Devoid of any wetness M9:Mouth feels tight ?
Time Frame: Prior to treatment on Day 8
Population: as for outcome 21
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants
  Q40: Strongly disagree | 6 | 8
  Q40: Disagree | 12 | 6
  Q40: Disagree a little | 3 | 4
  Q40: Agree a little | 15 | 11
  Q40: Agree | 11 | 11
  Q40: Strongly agree | 6 | 7
  Q41: Strongly disagree | 9 | 12
  Q41: Disagree | 20 | 9
  Q41: Disagree a little | 6 | 5
  Q41: Agree a little | 10 | 6
  Q41: Agree | 6 | 7
  Q41: Strongly agree | 2 | 8
  Q42: Strongly disagree | 10 | 9
  Q42: Disagree | 14 | 9
  Q42: Disagree a little | 8 | 6
  Q42: Agree a little | 10 | 8
  Q42: Agree | 5 | 8
  Q42: Strongly agree | 6 | 7
  Q43: Strongly disagree | 3 | 3
  Q43: Disagree | 4 | 1
  Q43: Disagree a little | 3 | 0
  Q43: Agree a little | 12 | 9
  Q43: Agree | 17 | 18
  Q43: Strongly agree | 14 | 16
  Q44: Strongly disagree | 3 | 4
  Q44: Disagree | 8 | 3
  Q44: Disagree a little | 9 | 4
  Q44: Agree a little | 8 | 13
  Q44: Agree | 18 | 16
  Q44: Strongly agree | 7 | 7
  Q45: Strongly disagree | 10 | 6
  Q45: Disagree | 16 | 12
  Q45: Disagree a little | 9 | 7
  Q45: Agree a little | 12 | 10
  Q45: Agree | 4 | 7
  Q45: Strongly agree | 2 | 5
  Q46: Excellent | 5 | 3
  Q46: Very Good | 20 | 14
  Q46: Good | 11 | 12
  Q46: Fair | 16 | 14
  Q46: Poor | 1 | 4
  QM1: Strongly disagree | 5 | 6
  QM1: Disagree | 15 | 5
  QM1: Disagree a little | 2 | 2
  QM1: Agree a little | 18 | 14
  QM1: Agree | 11 | 16
  QM1: Strongly agree | 2 | 4
  QM2: Strongly disagree | 7 | 10
  QM2: Disagree | 14 | 7
  QM2: Disagree a little | 6 | 5
  QM2: Agree a little | 18 | 9
  QM2: Agree | 8 | 13
  QM2: Strongly agree | 0 | 3
  QM3: Strongly disagree | 12 | 11
  QM3: Disagree | 17 | 10
  QM3: Disagree a little | 9 | 8
  QM3: Agree a little | 12 | 8
  QM3: Agree | 3 | 8
  QM3: Strongly agree | 0 | 2
  QM4: Strongly disagree | 8 | 3
  QM4: Disagree | 15 | 9
  QM4: Disagree a little | 8 | 5
  QM4: Agree a little | 17 | 12
  QM4: Agree | 4 | 14
  QM4: Strongly agree | 1 | 4
  QM5: Strongly disagree | 9 | 3
  QM5: Disagree | 14 | 10
  QM5: Disagree a little | 9 | 7
  QM5: Agree a little | 15 | 11
  QM5: Agree | 5 | 12
  QM5: Strongly agree | 1 | 4
  QM6: Strongly disagree | 5 | 4
  QM6: Disagree | 7 | 2
  QM6: Disagree a little | 6 | 1
  QM6: Agree a little | 23 | 16
  QM6: Agree | 9 | 13
  QM6: Strongly agree | 3 | 11
  QM7: Strongly disagree | 5 | 3
  QM7: Disagree | 10 | 1
  QM7: Disagree a little | 4 | 3
  QM7: Agree a little | 18 | 12
  QM7: Agree | 11 | 21
  QM7: Strongly agree | 5 | 7
  QM8: Strongly disagree | 7 | 3
  QM8: Disagree | 10 | 3
  QM8: Disagree a little | 7 | 4
  QM8: Agree a little | 15 | 11
  QM8: Agree | 12 | 21
  QM8: Strongly agree | 2 | 5
  QM9: Strongly disagree | 7 | 5
  QM9: Disagree | 16 | 4
  QM9: Disagree a little | 7 | 6
  QM9: Agree a little | 14 | 16
  QM9: Agree | 7 | 15
  QM9: Strongly agree | 2 | 1

31. Secondary Outcome: Mean Response to Post-Product Use Sensory Questionnaire (PPUSQ) on Day 1, Day 3, Day 8
Description: Participants answered 4 questions on PPUSQ as follows: Q1:Which of the following statements best describes how much you liked the product overall?(rated on scale of 1-6, 1=Did not like it at all; 2=Did not like it that much; 3=Like it slightly; 4=Like it somewhat; 5=Like it very much; 6=Like it extremely), Q2:How pleasant would you say the flavor of the product was?(rated on scale of 1-5, 1=Not pleasant at all; 2=Slightly pleasant; 3=Moderately pleasant; 4=Very pleasant; 5=Extremely pleasant), Q3:How gentle would you say the product was?(rated on a scale of 1-7, 1=Not gentle at all; 2=Barely gentle; 3=Slightly gentle; 4=Moderately gentle; 5=Very gentle; 6=Extremely gentle; 7=The most gentle product imaginable), Q4:How fresh would you say your mouth felt after using the product?(rated on a scale of 1-5; 1=Not at all fresh; 2=Not very fresh; 3=Somewhat fresh; 4=Very fresh; 5=Extremely fresh) & response to these questions was reported. Scale score was averaged to calculate the response
Time Frame: Day 1, Day 3, Day 8
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
score on a scale
  Day 1: Q1 | 4.60 (0.158) | 4.81 (0.168)
  Day 3: Q1 | 4.64 (0.161) | 4.53 (0.171)
  Day 8: Q1 | 4.75 (0.155) | 4.72 (0.164)
  Day 1: Q2 | 3.77 (0.172) | 3.54 (0.183)
  Day 3: Q2 | 3.67 (0.164) | 3.09 (0.174)
  Day 8: Q2 | 3.70 (0.167) | 3.53 (0.177)
  Day 1: Q3 | 5.21 (0.174) | 5.76 (0.184)
  Day 3: Q3 | 5.32 (0.158) | 5.86 (0.167)
  Day 8: Q3 | 5.24 (0.159) | 5.81 (0.169)
  Day 1: Q4 | 4.11 (0.152) | 3.38 (0.161)
  Day 3: Q4 | 3.93 (0.155) | 3.21 (0.165)
  Day 8: Q4 | 4.09 (0.150) | 3.20 (0.159)

32. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events on administration of investigational product from screening (Day 1) to 5 days after last administration of the product on Day 8. Number of participants with TEAEs were reported.
Time Frame: up to 13 days
Population: Analysis for this outcome was conducted on safety population which included all participants who were randomized and received at least one dose of study treatment during the study.
Measure: Number; unit: Number of participants
Arm/Group | Experimental Mouthwash | Mineral Water
Number analyzed (Participants) | 53 | 47
Number of participants | 12 | 4

ADVERSE EVENTS:
Time Frame: up to 13 days (from screening [Day 1] to 5 days after administration of last product on Day 8)
Arm/Group | Experimental Mouthwash | Mineral Water
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/47
Other Adverse Events (participants affected / at risk) | 12/53 | 4/47
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Mouthwash (N=53) | Mineral Water (N=47)
ORAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0
PARAESTHESIA ORAL (Gastrointestinal disorders) | 2 | 0
TONGUE COATED (Gastrointestinal disorders) | 1 | 1
GLOSSODYNIA (Gastrointestinal disorders) | 1 | 0
LIP DRY (Gastrointestinal disorders) | 1 | 0
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1
BURN ORAL CAVITY (Injury, poisoning and procedural complications) | 1 | 1
TONGUE INJURY (Injury, poisoning and procedural complications) | 2 | 0
LIP INJURY (Injury, poisoning and procedural complications) | 1 | 0
MOUTH INJURY (Injury, poisoning and procedural complications) | 1 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 1
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.